CLINICAL TRIAL: NCT03746496
Title: Point-of-care Analyses of Intraosseous Blood Samples Within Critically Ill Patients
Brief Title: POC Analysis of IO Blood Samples Within Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: FinnHEMS Oy (Unknown)
Responsible Party: Principal Investigator, Jouni Nurmi, MD, Docent, Helsinki University Central Hospital
Other Study IDs: 1234567890
Record Dates: First submitted 2018-09-27; First posted 2018-11-19 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Critically Ill
Keywords: intraosseous; blood gas analysis; emergency medicine; critically ill; point-of-care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pre-hospital emergency patients: Patient in a need of an IO-access. Patient in a need of point-of-care laboratory analysis. Over 18 years. Alive (no Cardiac arrest.)
  Interventions: Diagnostic Test: point-of-care laboratory analysis

INTERVENTIONS:
Diagnostic Test: point-of-care laboratory analysis — POC analysis with i-STAT POC analyser from the intraosseous and arterial blood

SUMMARY:
This study aims to investigate whether point-of-care (POC) analysis of intraosseous (IO) blood samples from critically ill emergency patients are accurate enough for emergency decision making, in comparison with arterial point-of-care samples.

DETAILED DESCRIPTION:
Intravenous access is sometimes difficult to achieve due to vasoconstriction or centralization of circulation. Feasible IO-access with power-driven device is a standard alternative method of vascular access for critically ill patients. It is still unclear whether results of IO samples agree with venous or arterial blood samples so that they could be used in clinical decision-making.

After intraosseous access has been established for fluid resuscitation or medication, a common practice is to aspirate a small amount of blood to verify the proper location of the IO-needle.

POC-testing can provide emergency physicians or paramedics with important information about the patients. Could bone marrow samples be used for POC-testing instead of arterial or venous blood for emergency treatment decision-making or patient allocation?

Several animal and human studies have been published to investigate the correlation between IO versus venous or arterial blood values. Investigators of this study have performed a study in healthy volunteers and discovered that there is a good agreement for some laboratory parameters (pH, gluc, lact), but for K the agreement is poor. Our study group has as well performed a study in critically ill animals investigating the agreement during cardiac arrest and resuscitation. Te evidence about critically ill people is still week.

Aim of this study is to analyze the reliability of analysis of IO samples compared to arterial blood samples within critically ill adult emergency patients.

The hypotheses of this study are:

1. Principally, it is possible to analyze IO blood samples with a POC device.
2. The results are reliable enough to guide emergency treatment.

If both hypotheses prove to be true, the method can be immediately used in emergency medical situations, e.g. in searching for reversible causes of cardiac arrest.

Setting

Prospective, observational study with 35 prehospital emergency patients. The IO-samples are collected from the small amount of blood, which is aspirated from intraosseous space to confirm the correct needle placement. The IO needles are inserted to the patients for emergency treatment, not because of the study. Critically ill patients, to whom emergency doctors are inserting an intraosseous needle for emergency fluid or drug treatment, are included in the study.

Samples will be analyzed by using an i-STAT point of care analyzer (i-STAT® handheld, Abbot Point of Care Inc. U.S.A) using CG8+ cartridges to analyse Hb, Na, K, pH, pCO2, pO2, TCO2, HCO3, BE, and SpO2. The reliability of the results comparing the IO and arterial samples will be tested with Bland-Altman method by calculating the bias with 95% confidence intervals.

Ethical issues

The ethical committee of Medical Faculty of University of Helsinki has approved the research. Informed consent is waived.

Time plan

The samples will be collected during years 2017 - 2019. The analysis will be performed in the end of the year 2019.

ELIGIBILITY:
Inclusion Criteria:

* need for point-of-care analysis
* need for intraosseous access

Exclusion Criteria:

* cardiac arrest
* ability to understand the consent issues in Finnish, Swedish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency patients, which are met by the helicopter emergency unit during their normal tasks
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
agreement between intraosseous (IO) and arterial POC analyses | Samples are analysed immediately after the sample has been taken. Statistical analysis about the agreement performed when the whole data has been collected.
  agreement analysed with Bland-Altman method from IO and arterial blood samples, which have been analysed with iSTAT point-of care analyser for following parameters: Hb, pH, BE, HCO3, pO2, pCO2, glucose, Na, K, iCa

CONTACTS AND LOCATIONS:
Overall Officials: Jouni Nurmi, M.D. Ph D, Principal Investigator — University of Helsinki, Helsinki University hospital
Locations (1):
- FinnHEMS10, Emergency Medicine and Services, Helsinki University Hospital, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jousi M, Laukkanen-Nevala P, Nurmi J. Analysing blood from intraosseous access: a systematic review. Eur J Emerg Med. 2019 Apr;26(2):77-85. doi: 10.1097/MEJ.0000000000000569. PMID 30124518
- [Result] Jousi M, Saikko S, Nurmi J. Intraosseous blood samples for point-of-care analysis: agreement between intraosseous and arterial analyses. Scand J Trauma Resusc Emerg Med. 2017 Sep 11;25(1):92. doi: 10.1186/s13049-017-0435-4. PMID 28893316
- [Result] Backman S, Angerman-Haasmaa S, Jousi M, Siitonen S, Salmela K. ABO and D typing and alloantibody screening in marrow samples: relevance to intraosseous blood transfusion. Transfusion. 2018 Jun;58(6):1372-1376. doi: 10.1111/trf.14557. Epub 2018 Mar 1. PMID 29492974
- [Result] Tallman CI, Darracq M, Young M. Analysis of intraosseous blood samples using an EPOC point of care analyzer during resuscitation. Am J Emerg Med. 2017 Mar;35(3):499-501. doi: 10.1016/j.ajem.2016.12.005. Epub 2016 Dec 12. PMID 27998615
- [Result] Veldhoen ES, de Vooght KM, Slieker MG, Versluys AB, Turner NM. Analysis of bloodgas, electrolytes and glucose from intraosseous samples using an i-STAT((R)) point-of-care analyser. Resuscitation. 2014 Mar;85(3):359-63. doi: 10.1016/j.resuscitation.2013.12.002. Epub 2013 Dec 31. PMID 24389357